CLINICAL TRIAL: NCT02617420
Title: Monitoring Adherence Using Mobile Technology
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0211
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intervention: All patients will be enrolled in one arm. These patients will have monitoring devices placed on their asthma controller and rescue medication, with data transmitted both to their smartphones and a dashboard accessed by their primary pediatric pulmonary provider.
  Interventions: Device: Propeller Health Monitoring Device

INTERVENTIONS:
Device: Propeller Health Monitoring Device

SUMMARY:
This study plans to learn more about how children use their asthma medicines. The investigators would like to see if special electronic monitoring devices that connect to smartphones and computers can help children to better manage their asthma

ELIGIBILITY:
Inclusion Criteria:

* age 6-17 years and their parents
* either 2 emergency department visits/prednisone bursts in the last 12 months or at least 1 asthma related hospitalization in the last 12 months
* requiring daily controller therapy with either inhaled corticosteroids or combination corticosteroids/long acting beta agonist (LABA).
* Patients using metered dose inhaler therapy would be eligible. Patients may also be on leukotriene antagonists,
* Must be made aware that they will have to read and accept to the terms of the User Agreement prior to enrollment in the study. If they do not agree they will not be able to continue participation. The User agreement will be read agreed to electronically when they begin using the device, however a paper version will be provided at the time of consent upon request.

Exclusion Criteria:

* Primary language other than English or Spanish
* Presence of other significant chronic lung disease including cystic fibrosis, interstitial lung disease, tracheostomy status.
* Patients using diskus therapy.
* Patients only on leukotriene antagonists.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study subjects would be drawn from the list of high risk asthma patients and by pre-clinic chart review done by study investigator.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patient participants that rate the devices as easy to use | 3 months
  Measuring the feasibility and acceptability of monitoring devices for children ages 6-17 who are at high risk for asthma exacerbation, by having children use the devices and having children/parents answer survey questions regarding their impressions of the product at the beginning of use and after 1.5 and 3 months of use.
Number of provider participants that rate the devices as easy to use | 3 months
  Measuring the feasibility and acceptability of monitoring devices for children ages 6-17 who are at high risk for asthma exacerbation, by having children use the devices and having providers answer survey questions regarding their impressions of the product at the beginning of use and after 1.5 and 3 months of use.

SECONDARY OUTCOMES:
Number of patients/parents that exhibit behavioral changes with respect to taking asthma medications as a result of information gained from the monitoring devices. | 3 months
  How many parents/patients of high risk asthmatic children change behavior regarding how they administer their medications as a result of information that they gained from the devices regarding their adherence to their treatment regimen, gained via phone surveys at 1.5 and 3 months after using the devices. Patients are surveyed if children are greater than 12 years old. Parents are surveyed if children are 6-12 years old.
Number of pediatric pulmonary providers that exhibit behavioral changes with respect to prescribing asthma medications as a result of information gained from the monitoring devices. | 3 months
  Number of healthcare providers (physicians, nurse practitioners and physician assistants) that feel that their decision-making is affected regarding medication regimens for asthma based on information that they receive on patient adherence from the devices based on survey data gathered at study entry and 3 months after initiation of the devices will be measured.
Correlation of lung function to percent use of controller medications as measured by adherence devices. | 3 months
  Evaluate correlation of markers of lung function (spirometry, fractional exhaled nitric oxide (FeNO), with percent adherence as measured by the monitoring devices.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Szefler, MD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Derived] Hoch H, Kempe A, Brinton J, Szefler S. Feasibility of medication monitoring sensors in high risk asthmatic children. J Asthma. 2019 Mar;56(3):270-272. doi: 10.1080/02770903.2018.1446979. Epub 2018 Apr 11. No abstract available. PMID 29641374